CLINICAL TRIAL: NCT02511327
Title: Pertussis Immunization During Pregnancy: Assessment of the Role of Maternal Antibodies on Immune Responses in Term and Preterm Infants: the MAMA Study
Brief Title: Pertussis Immunization During Pregnancy: Effect in Term and Preterm Infants
Acronym: MAMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); Université Libre de Bruxelles (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Elke Leuridan, MD, PhD, Elke Leuridan, MD, PhD, Universiteit Antwerpen
Other Study IDs: cev003
Record Dates: First submitted 2015-07-22; First posted 2015-07-30 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Pertussis
Keywords: Pertussis; Pregnancy; Vaccination; Preterm; Breast milk; Humoral immune response; Cellular immune response; Maternal antibodies
MeSH Terms: conditions — Whooping Cough; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and breast milk samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Preterm born infants of vaccinated women: Preterm born infants (< 37 weeks of gestation) whose mothers have received an acellular pertussis vaccine during pregnancy, within the national recommended vaccination programme. Infant vaccination against pertussis is performed according to the national recommended schedule.
  Interventions: Drug: Infant pertussis vaccination
- Term born infants vaccinated women: Term born infants (>= 37 weeks of gestation) whose mothers have received an acellular pertussis vaccine during pregnancy, within the national recommended vaccination programme. Infant vaccination against pertussis is performed according to the national recommended schedule.
  Interventions: Drug: Infant pertussis vaccination
- Term born infants unvaccinated women: Term born infants (>= 37 weeks of gestation) whose mothers have not received an acellular pertussis vaccine during pregnancy. Infant vaccination against pertussis is performed according to the national recommended schedule.
  Interventions: Drug: Infant pertussis vaccination
- Preterm born infants unvaccinated women: Preterm born infants (< 37 weeks of gestation) whose mothers have not received an acellular pertussis vaccine during pregnancy.Infant vaccination against pertussis is performed according to the national recommended schedule.
  Interventions: Drug: Infant pertussis vaccination

INTERVENTIONS:
Drug: Infant pertussis vaccination — Infants receive pertussis vaccines according to the national recommended schedule
  Other Names: Infant pertussis containing vaccination

SUMMARY:
Young infants are most vulnerable to severe disease and even death when infected with Bordetella Pertussis. The current vaccines and vaccination programs do not guarantee protection of neonates. During the last weeks of pregnancy, maternal IgG antibodies are transferred actively to the fetus. Administration of a pertussis containing vaccine during pregnancy offers protection through high titers of maternal antibodies transferred to the child. Since transplacental transport is immature, infants who are born prior to 37 weeks of gestation, might be vulnerable to pertussis infection even though maternal vaccination was administered, but specific data are lacking. The primary aim of this observational study is to measure whether vaccination during pregnancy offers protection to preterm born infants through higher titers of maternal antibodies, despite immature transplacental transport. Four cohorts of mother-infant pairs will be recruited: term versus preterm born infants, born from either vaccinated women or not vaccinated women. These mother-infant pairs are recruited according to the vaccination status of the mother and to the gestational age at delivery. Pertussis specific antibody titers (anti-Pertussis Toxin, anti-Filamentous haemagglutinin, anti-Pertactin titers) will be monitored in blood samples of the mothers at delivery to measure the possible influence of both gestational age and maternal vaccination status. In order to measure the decline of maternal antibodies in the first weeks of life, blood will be taken from cords as well as from infants at 8 weeks of age, before the first infant pertussis vaccine is administered.

Pertussis antibodies to the same antigens will be measured in all infants after a primary series of acellular pertussis vaccines administered at 8,12 and 16 weeks of age and before and after a booster dose in the second year of life.

In addition, cellular mediated immune responses will be evaluated in a subgroup of infants before and after a primary series of infants vaccines. A last goal is to measure whether vaccination during pregnancy could offer additional maternal antibodies through breast milk. Again a comparison is made between preterm and term born infants, born from either vaccinated or unvaccinated women. The amount of lactoferrin and pertussis toxin specific IgA in breast milk samples will be measured in samples taken at birth (colostrum), and at several time points afterwards as long as breastfeeding is continued.

ELIGIBILITY:
Inclusion Criteria for participating women:

* Pregnancy
* Signed informed consent
* Intend to be available for follow-up visits and phone call access through 16 months following delivery
* Willing to have infant immunized with hexavalent vaccine according to the recommended Belgian schedule

Exclusion Criteria for participating women:

* Significant mental illness (e.g. schizophrenia, psychosis, major depression)
* Serious underlying immunological condition (e.g. immunosuppressive disease or therapy, human immunodeficiency virus (HIV) infection)
* Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk
* Receipt of a blood product or experimental medicine within 4 weeks prior to delivery
* Multiple pregnancies

Exclusion Criteria for children:

* No signed informed consent from both parents
* Severe reactions to any vaccine
* Serious underlying medical condition (e.g., genetic disorder (eg Down syndrome), immunosuppressive disease or therapy, human immunodeficiency virus (HIV) infection, lung/heart disease, liver/kidney disease, chronic or recurrent infections)
* Children suffering from primary humoral immune disorders (B cell related): severe X linked agammaglobulinaemia, CVID (Common variable immunodeficiency, late onset agammaglobulnaemia) and SAD (specific antibody deficiency); suffering from primary cellular immune deficiencies (T cell related): SCID (Severe combined immune deficiency syndrome), CID, hyper IGM syndrome, di George's syndrome and others; suffering from disorders in phagocytosis and chemotaxis (CGD, Schwach Diamond syndrome) and disorders from the complement cascade
* In addition children with oncologic disorders will be excluded. All these children can receive the inactivated pertussis vaccines, but will respond different from the normal population to vaccination.
* Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk.

Ages: 0 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Four cohorts of women-infant pairs will be recruited before or directly after delivery.
  A cohort of preterm born infants will be compared to term born infants, and both will be compared within groups of vaccinated women (adult acellular pertussis containing vaccine) or unvaccinated women.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Titers of maternal pertussis specific antibodies | From birth until 8 weeks of age
  Anti-Pertussis Toxin, anti-Filamentous Haemagglutinin and anti-pertactin immunoglobulin IgG titers, measured in blood samples taken from cord and at week 8 postpartum in all participating infants

SECONDARY OUTCOMES:
Titers of pertussis specific antibodies in infants after 3 doses of a pertussis vaccine | At the age of 5 months
  Anti-Pertussis Toxin, anti-Filamentous Haemagglutinin and anti-pertactin immunoglobulin IgG titers, measured in blood samples taken at 5 months (after a primary series of 3 vaccines)
Titers of pertussis specific antibodies in infants before and after a fourth dose of a pertussis vaccine | From 13 to 16 months
  Anti-Pertussis Toxin, anti-Filamentous Haemagglutinin and anti-pertactin immunoglobulin IgG titers, measured in blood samples taken before and 1 month after a fourth pertussis vaccine
Titers of pertussis specific antibodies in infants in-between the fourth and fifth dose of a pertussis vaccine | Around 3 years of age
  Anti-Pertussis Toxin, anti-Filamentous Haemagglutinin and anti-pertactin immunoglobulin IgG titers, measured in blood samples taken before and 1 month after a fourth pertussis vaccine
Titers of pertussis specific antibodies in infants before and after a fifth dose of a pertussis vaccine | From 5 to 6 years of age
  Anti-Pertussis Toxin, anti-Filamentous Haemagglutinin and anti-pertactin immunoglobulin IgG titers, measured in blood samples taken before and 1 month after a fourth pertussis vaccine
Th1 immune responses in preterm and term born infants before and after a primary series of infant pertussis vaccines | From 8 weeks of age until 16 months of age
  Measurement of Th1 markers in a convenience sample of infants after primary and booster pertussis vaccination
Th2 immune responses in preterm and term born infants before and after a primary series of infant pertussis vaccines | From 8 weeks of age until 16 months of age
  Measurement of Th2 markers in a convenience sample of infants after primary and booster pertussis vaccination
Th1 & Th2 immune responses in preterm and term born infants before and after a fifth booster dose of a pertussis vaccine | From 5 to 6 years of age
  Measurement of Th1 and Th2 markers in a convenience sample of infants before and after a pertussis booster vaccination
Titers of pertussis specific IgA antibodies in breast milk | From birth until 3 months postpartum
  Measurement of anti-Pertussis Toxin IgA, total IgA and lactoferrin titers in breast milk samples taken at birth, at week 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Elke Leuridan, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Embacher S, Maertens K, Herzog SA. Half-life Estimation of Pertussis-Specific Maternal Antibodies in (Pre)Term Infants After In-Pregnancy Tetanus, Diphtheria, Acellular Pertussis Vaccination. J Infect Dis. 2023 Nov 28;228(11):1640-1648. doi: 10.1093/infdis/jiad212. PMID 37285482
- [Derived] Maertens K, Orije MRP, Huoi C, Boisnard F, Lyabis O. Immunogenicity of a liquid hexavalent DTaP-IPV-HB-PRP approximately T vaccine after primary and booster vaccination of term and preterm infants born to women vaccinated with Tdap during pregnancy. Vaccine. 2023 Jan 16;41(3):795-804. doi: 10.1016/j.vaccine.2022.12.021. Epub 2022 Dec 15. PMID 36528443
- [Derived] Orije MRP, Garcia-Fogeda I, Van Dyck W, Corbiere V, Mascart F, Mahieu L, Hens N, Van Damme P, Cools N, Ogunjimi B, Maertens K, Leuridan E. Impact of Maternal Pertussis Antibodies on the Infants' Cellular Immune Responses. Clin Infect Dis. 2022 Aug 31;75(3):442-452. doi: 10.1093/cid/ciab972. PMID 34849638
- [Derived] Maertens K, Orije MRP, Herzog SA, Mahieu LM, Hens N, Van Damme P, Leuridan E. Pertussis Immunization During Pregnancy: Assessment of the Role of Maternal Antibodies on Immune Responses in Term and Preterm-Born Infants. Clin Infect Dis. 2022 Jan 29;74(2):189-198. doi: 10.1093/cid/ciab424. PMID 33971009
- [Derived] Orije MRP, Lariviere Y, Herzog SA, Mahieu LM, Van Damme P, Leuridan E, Maertens K. Breast Milk Antibody Levels in Tdap-Vaccinated Women After Preterm Delivery. Clin Infect Dis. 2021 Sep 15;73(6):e1305-e1313. doi: 10.1093/cid/ciab260. PMID 33768227